CLINICAL TRIAL: NCT06881173
Title: Efficacy of Meridian Energy and Heart Rate Variability in Patients with Ocular Myasthenia Gravis by Using Chinese and Western Medicine Treatment
Brief Title: The Effectiveness of Bu Zhong Yi Qi Tang in Patients with Myasthenia Gravis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng, yu-ting (Other)
Responsible Party: Sponsor-Investigator, Cheng, yu-ting, Principal Investigator, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220305R
Record Dates: First submitted 2024-08-06; First posted 2025-03-18 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-08

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — bu-zhong-yi-qi-tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Have taken Bu Zhong Yi Qi Tang
  Interventions: Drug: Bu Zhong Yi Qi Tang
- control group (Placebo Comparator): Have taken caramel dyed starch placebo
  Interventions: Drug: caramel dyed starch placebo

INTERVENTIONS:
Drug: Bu Zhong Yi Qi Tang — The experimental group took 15g of Buzhong Yiqi Decoction concentrated powder, 3 times a day, 1 packet each time.
  Other Names: TE202208013
  Arms: Experimental group
Drug: caramel dyed starch placebo — The control group took 15 grams of caramel dyed starch placebo, 1 pack at a time, 3 times a day.
  Other Names: starch placebo
  Arms: control group

SUMMARY:
Research Background: According to the Myasthenia Gravis Foundation of America (MGFA, 2015), the estimated prevalence of myasthenia gravis is 14-20 per 100,000 people, with a higher prevalence in young female individuals compared to males. However, as individuals age, especially after the age of 50, the prevalence in males becomes higher than in females. myasthenia gravis patients often experience varying degrees of disability, leading to the need for long-term medical care, medication, and lifestyle adjustments. This also gives rise to subsequent challenges in caregiving, affecting both the patients' families and society.

DETAILED DESCRIPTION:
:This study aims to assess the effectiveness of using a combination of traditional Chinese and Western medicine,to improve the meridian energy and autonomic nervous system function of myasthenia gravis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ocular myasthenia by a doctor
* Western medicine prescriptions only take oral Mestinon (Pyrido stigmine Bromide)
* Patients over 20 years old
* Can understand and understand Those who can speak Mandarin or Taiwanese
* those with a clear state of consciousness and no diagnosis of mental illness
* patients and their families who are willing to receive precise integrated treatment of traditional Chinese and Western medicine.

Exclusion Criteria:

* Patients with liver failure or kidney failure
* Allergy symptoms to traditional Chinese medicine, such as skin itching and redness
* Patients with malignant tumors
* Patients currently undergoing radiotherapy and chemotherapy
* Pregnant
* Cardiac rhythm device implementer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
meridian energy | 12 weeks
  After taking Buzhong Yiqi Decoction, the energy of the meridians can be balanced. Use a meridian measuring instrument to measure the meridians of the whole body and improve the energy of the meridians to the range of 40-60.
autonomic nervous system function | 12 weeks
  After taking Buzhong Yiqi Decoction, it can change the autonomic nervous system (ANS), reduce the sympathetic nerve energy, increase the parasympathetic nerve energy, and set the standard value of the autonomic nervous system activity between 40-60

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Han Liu, Study Chair — project leader
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No